CLINICAL TRIAL: NCT00539240
Title: Role of Pain Modulation in GERD Patients Who Failed Standard Dose PPI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-022-04F
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: acid reflux; acid regurgitation; esophagitis; GERD; heartburn; pain; peptic
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis; Heartburn; Pain | interventions — Rabeprazole; Nortriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rabeprazole morning/evening placebo bedtime (Placebo Comparator): AciPhex 20 mg BID and once daily placebo
  Interventions: Drug: Rabeprazole 20 mg two times, Placebo at bedtime
- Rabeprazole breakfast, placebo dinner and bedtime (Placebo Comparator): AcipHex 20 mg once daily and BID placebo
  Interventions: Drug: Rabeprazole 20mg, placebo dinner and bedtime
- Rabeprazole breakfast, placebo dinner, nortriptyline bedtime (Active Comparator): AcipHex 20 mg once daily, placebo once daily and nortriptyline once daily
  Interventions: Drug: Rabeprazole 20mg,placebo dinner ,Low dose Tricyclic Antidepressant

INTERVENTIONS:
Drug: Rabeprazole 20mg, placebo dinner and bedtime — Breakfast study medication - Rabeprazole 20mg, matching placebo at dinner , Placebo for tricyclic antidepressant at bedtime
  Other Names: AcipHex
  Arms: Rabeprazole breakfast, placebo dinner and bedtime
Drug: Rabeprazole 20 mg two times, Placebo at bedtime — Breakfast & Dinner study medication - Rabeprazole, placebo for tricyclic antidepressant at bedtime
  Other Names: Aciphex
  Arms: Rabeprazole morning/evening placebo bedtime
Drug: Rabeprazole 20mg,placebo dinner ,Low dose Tricyclic Antidepressant — Rabeprazole (Breakfast) study medication, dinner placebo medication, tricyclic antidepressant at bedtime
  Other Names: Nortriptyline and Aciphex
  Arms: Rabeprazole breakfast, placebo dinner, nortriptyline bedtime

SUMMARY:
The purpose of this project is to compare the efficacy (how successful) 1) standard-dose proton pump inhibitor (PPI) (rabeprazole 20 mg once daily) (a medication that completely blocks the stomach from producing acid) plus low dose tricyclic antidepressant (nortriptyline 50mg) (TCA); 2) double-dose PPI (rabeprazole 20 mg twice a day); to 3) standard-dose PPI (rabeprazole 20mg once daily) and placebo (an inactive substance, like a sugar pill) to determine the relative symptom resolution and health-related quality of life in gastroesophageal reflux disease (a disease characterized by a burning sensation (heartburn) behind the breast bone caused by a backflow of stomach contents into the esophagus) (GERD) patients who fail standard-dose PPI and you will be randomly assigned (similar to flipping a coin) to one of the three groups.

DETAILED DESCRIPTION:
Failure of standard dose PPI to control GERD symptoms has been increasingly encountered in clinical practice (both primary care and sub-specialties) and has become one of the most challenging therapeutic dilemmas in GERD management. It has been estimated that up to 30% of the patients receiving PPI once daily will continue to report typical GERD symptoms [1]. Presently, increasing the PPI dose has been the standard of care in these patients [2]. However, success in relieving refractory GERD symptoms with such a therapeutic approach has been extremely limited, resulting in frustration of both the patient as well as the health care provided. Furthermore, patients who fail PPI will continue to seek medical attention and may undergo a variety of invasive or non-invasive tests, and thus consume already limited health care resources. Recent advancement in the understanding of the diverse composition of the different GERD groups as well as symptom generation has led to the recognition of alteration in pain perception as an important contributing factor for PPI failure in some and the presence of non-acid related stimuli in others [3].

This study will clarify for the first time the role of pain modulation in patients who failed standard dose of PPI. The clinical experience with doubling the PPI dose, which is the current standard of care, has been very limited and relatively disappointing. Additionally, this study may identify the group of PPI failure patients that may benefit from doubling the dose of PPI and the group that will benefit more from adding a pain modulator. This study is timely, has never been performed and addresses a prevalent emerging clinical dilemma in GI as well as primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated with a PPI, but continue to experience GERD symptoms (such as heartburn) at least 2 times per week.

Exclusion Criteria:

* Known allergy or intolerance to TCA
* History of serious arrhythmia or use of anti-arrhythmics
* History of seizures
* Subjects with significant co-morbidity, e.g., cardiovascular, respiratory, urogenital, renal, gastrointestinal, hepatic, hematological, endocrine, neurologic or psychiatric
* With evidence or history of drug abuse within the past 6 months
* Erosive esophagitis, esophageal ulceration, peptic stricture, Barrett's esophagus or adenocarcinoma of the esophagus on endoscopy
* History of esophagogastric surgery
* Gastric or duodenal lesions (ulcer, tumor, etc.)
* Women who are pregnant or of childbearing age who are not on contraception
* Patients who are unwilling or unable to provide informed consent
* Insulin dependent diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2006-04; Primary Completion 2010-04 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Arizona VA Health Care System, Tucson, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from GI clinic in VA medical center between 4/19/2006 and 3/31/2010
Pre-assignment Details: Eligibility screening occurred prior to randomization. Of 236 patients enrolled, 68 patients were not randomized due to abnormal endoscopy (14 patients), asymptomatic during run-in period (2 patients), lost to follow-up (11 patients), consent withdrawal, protocol deviation and screen failure (32 patients) and other causes (9 patients).
Groups:
- Arm 1: AciPhex 20 mg BID and once daily placebo
  Rabeprazole 20mg, placebo dinner and bedtime: Breakfast study medication - Rabeprazole 20mg, matching placebo at dinner , Placebo for tricyclic antidepressant at bedtime
- Arm 2: AcipHex 20 mg once daily and BID placebo
  Rabeprazole 20 mg two times, Placebo at bedtime: Breakfast & Dinner study medication - Rabeprazole, placebo for tricyclic antidepressant at bedtime
- Arm 3: AcipHex 20 mg once daily, placebo once daily and nortriptyline once daily
  Rabeprazole 20mg,placebo dinner ,Low dose Tricyclic Antidepressant: Rabeprazole (Breakfast) study medication, dinner placebo medication, tricyclic antidepressant at bedtime
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 59 | 55 | 54
Completed | 53 | 48 | 39
Not Completed | 6 | 7 | 15
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Adverse Event | 3 | 1 | 10

BASELINE CHARACTERISTICS:
Population: Number of randomized subjects
Groups:
- AciPhex 20 mg BID and Once Daily Placebo: AciPhex 20 mg BID and once daily placebo
  Rabeprazole 20mg, placebo dinner and bedtime: Breakfast study medication - Rabeprazole 20mg, matching placebo at dinner , Placebo for tricyclic antidepressant at bedtime
- AcipHex 20 mg Once Daily and BID Placebo: AcipHex 20 mg once daily and BID placebo
  Rabeprazole 20 mg two times, Placebo at bedtime: Breakfast & Dinner study medication - Rabeprazole, placebo for tricyclic antidepressant at bedtime
- AcipHex 20 mg Once, Placebo Once, Nortriptyline: AcipHex 20 mg once daily, placebo once daily and nortriptyline once daily
  Rabeprazole 20mg,placebo dinner ,Low dose Tricyclic Antidepressant: Rabeprazole (Breakfast) study medication, dinner placebo medication, tricyclic antidepressant at bedtime
- Total: Total of all reporting groups
Arm/Group | AciPhex 20 mg BID and Once Daily Placebo | AcipHex 20 mg Once Daily and BID Placebo | AcipHex 20 mg Once, Placebo Once, Nortriptyline | Total
Number analyzed (Participants) | 59 | 55 | 54 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13.8) | 54.8 (13.4) | 56 (11.5) | 55.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 13 | 48
  Male | 43 | 36 | 41 | 120
Region of Enrollment [Number; unit: participants]
  United States | 59 | 55 | 54 | 168
Body Mass Index [Mean (Standard Deviation); unit: kg/meter-squared] | 29.4 (6.1) | 29.3 (6.5) | 29.8 (4.6) | 29.5 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Daytime Heartburn, Number of Days in Week Symptoms Intensity Score < 3 (Better)
Description: the number of days with Symptom Intensity Score < 3 (better) for daytime heartburn during week 6 as compared to baseline
Time Frame: Symptom control after 6 weeks of treatment
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 53 | 48 | 39
days | 6.6 (0.9) | 5.9 (2.2) | 6.1 (1.8)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = 0.04, Regression, Linear — P<0.05 considered statistically significant. No adjustment for multiple comparisons; adjusted for age, sex, BMI and ethnicity
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; Test type: Superiority or Other; p = 0.50, Regression, Linear — P<0.05 considered statistically significant, No adjustment for multiple comparisons; adjusted for age, sex, BMI and ethnicity

2. Secondary Outcome: Health Related Quality of Life
Description: SF-36 Physical Component Score (higher number better quality of life), is a measure of overall physical quality of life distinct from mental health. The range is 0 - 100. It has been adjusted to US national norms so that a score of 50 corresponds to the national mean.
Time Frame: end of study
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 53 | 48 | 39
units on a scale | 42.0 (10.3) | 37.7 (11.0) | 37.7 (11.0)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3; Test type: Superiority or Other; p = 0.19, ANCOVA — P<0.05 considered statistically significant. No adjustment for multiple comparisons (no post-hoc contrasts performed); Adjusted for baseline score and personality traits (SCL-90)

3. Primary Outcome: Nighttime Heartburn, Number of Days in Week Symptom Activity Score <3 (Better) in Week 6 Compared to Baseline
Description: the number of days with Symptom Intensity Score < 3 (better) for nighttime heartburn during week 6 as compared to baseline
Time Frame: Symptom control after 6 weeks of treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 53 | 48 | 39
days | 6.6 (0.9) | 5.8 (2.0) | 6.0 (1.6)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = 0.04, Regression, Linear — P<0.05 considered statistically significant, No adjustment for multiple comparisons; adjusted for age, sex, BMI and ethnicity
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; Test type: Superiority or Other; p = 0.50, Regression, Linear — P<0.05 considered statistically significant, no adjustment for multiple comparisons; adjusted for age, sex, BMI and ethnicity

4. Primary Outcome: Acid Regurgitation, Number of Days in Week Symptoms Intensity Score < 3 (Better)
Description: the number of days with Symptom Intensity Score < 3 (better) for acid regurgitation during week 6 as compared to baseline
Time Frame: Symptom control after 6 weeks of treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 53 | 48 | 39
days | 6.7 (0.8) | 5.9 (2.1) | 6.3 (1.4)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = 0.04, Regression, Linear — P<0.05 considered statistically significant. No adjustment for multiple comparisons; adjusted for age, sex, BMI and ethnicity
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; Test type: Superiority or Other; p = 0.20, Regression, Linear — P<0.05 considered statistically significant. No adjustment for multiple comparisons; adjusted for age, sex, BMI and ethnicity

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 3/59 | 1/55 | 10/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=59) | Arm 2 (N=55) | Arm 3 (N=54)
Flu like symptoms (General disorders) | 0 | 1 | 0
skin ulceration (Gastrointestinal disorders) | 1 | 0 | 0 — ulcer on tongue
Other, Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Rash (type unspecified) on face
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 — "Stomach cramps"
Somnolence (Nervous system disorders) | 1 | 0 | 3 — "Drowsiness"
Other, Renal and urinary disorders (Renal and urinary disorders) | 0 | 0 | 1 — "urinary difficulty" (type unspecified)
Flushing (Vascular disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Recruitment challenges, including difficulty finding patients who "fail" PPI but had not already been prescribed doubled dose. Necessitated a no-cost extension to complete recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No